CLINICAL TRIAL: NCT04330781
Title: Patient-reported Outcome After Radiotherapy of Oral Cavity and Sinonasal Cancer Using an Intraoral Stent
Brief Title: Radiotherapy of Head and Neck Cancer Using an Intraoral Stent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Einar Dale, Senior Consultant, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-38
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-12

CONDITIONS: Oral Cavity Cancer; Sinonasal Cancer
Keywords: Radiotherapy; Intraoral stent; Head and neck cancer; Patient-reported outcome
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): N=123
  Interventions: Device: Intraoral stent
- Control group (Active Comparator): N=31
  Interventions: Other: No intraoral stent

INTERVENTIONS:
Device: Intraoral stent — Radiotherapy with intraoral stent
  Arms: Intervention group
Other: No intraoral stent — Radiotherapy without intraoral stent
  Arms: Control group

SUMMARY:
Radiotherapy of oral cavity cancer and sinonasal cancer is associated with acute and late morbidity. Use of an intraoral stent will provide a larger distance between the tongue and palate and can reduce side-effects. The aim of the present study is to confirm that an intraoral stent is not a significant bother to the patients.

DETAILED DESCRIPTION:
The investigators have previously performed a pilot study on the feasibility of the intraoral stent in patients receiving radiotherapy for tongue cancer. It was found that most of the patients tolerated the stent. The mean radiation dose to the hard palate was reduced by 61% (absolute percentage) as compared with a control group not using the stent. Based on these results, the investigators wish to perform a study on a larger cohort to confirm that the intraoral stent will not lead to increased symptoms towards the end of the radiotherapy period.

ELIGIBILITY:
Inclusion Criteria:

* Radiation dose 30 Gy or higher
* Cancer in the inferior part of the oral cavity (e.g. tongue or floor of mouth cancer) or superior part of the oral cavity (e.g. hard palate) or sinonasal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Ability to understand and answer questionnaire

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Patient-reported outcome | At the end of radiotherapy (5-6 weeks)
  Less than 10% change (non-inferiority) in sum of pain scores (no 31-34) in questionnaire European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - H&N 35 plus 3 extra questions regarding pain in the palate, tongue and lips

CONTACTS AND LOCATIONS:
Overall Officials: Einar Dale, MD PhD, Principal Investigator — Senior Consultant
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bø B, Furre T, Dale E. Radiotherapy of tongue cancer using an intraoral stent: a pilot study. Journal of Radiotherapy in Practice. 2021;21(3):370-6.